CLINICAL TRIAL: NCT06925867
Title: A Frequency-Modulated Music Intervention to Enhance Cognitive Processing Therapy (CPT) for PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Wright-Patterson Air Force Base (Unknown)
Responsible Party: Principal Investigator, Jacek Kolacz, Research Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024H0212; HT94252410126 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: music; hyperarousal; cognitive processing therapy
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frequency Filtered Music (Experimental): Participants will receive 10 daily sessions of cognitive processing therapy (2 weeks total) and listen to 15 minutes of frequency filtered classical music before each therapy session (2.5 hours music listening total).
  Interventions: Other: Frequency Filtered Music; Behavioral: Cognitive Processing Therapy for PTSD
- Unfiltered Music (Active Comparator): Participants will receive 10 daily sessions of cognitive processing therapy (2 weeks total) and listen to 15 minutes of classical music with no frequency filtering before each therapy session (2.5 hours music listening total).
  Interventions: Other: Unfiltered Music; Behavioral: Cognitive Processing Therapy for PTSD

INTERVENTIONS:
Other: Frequency Filtered Music — The frequency filtered music intervention is 2.5 hours of classical music that has been filtered by applying an algorithm to alternate narrowing and expanding the range of acoustic frequencies over time, with the alternations intensifying in frequency range over the course of administration. The filtering is optimized for the frequency response of adult human hearing and intended to mimic the expression of the human voice around a central set of frequencies of 800-1200 Hz, the approximate resonant frequency of the human ear. The filtering method is similar to adjusting the treble and bass settings on a stereo system while music is playing; the melody and instruments can still be heard, but the highest and lowest pitches are modulated over time.
  Other Names: Safe and Sound Protocol
  Arms: Frequency Filtered Music
Other: Unfiltered Music — The unfiltered music intervention is 2.5 hours of classical music with. The playlist of pieces is identical to the filtered music condition.
  Arms: Unfiltered Music
Behavioral: Cognitive Processing Therapy for PTSD — Cognitive processing therapy (CPT) is a cognitive therapy that focuses on why patients believe the traumatic event occurred, how that event affected their beliefs about self and others, and how to evaluate their beliefs. Patients then learn to label events, thoughts, and subsequent emotions while the therapist helps them examine the facts and context of the trauma through Socratic questioning. Using progressive worksheets, patients are taught to examine their own thoughts and emotions and develop new, more balanced thinking about traumatic events.

SUMMARY:
The goal of this clinical trial is to learn if the addition of frequency filtered music (Safe and Sound Protocol) to daily cognitive processing therapy improves effectiveness for reducing PTSD symptoms. The main questions it aims to answer are:

* Does the addition of frequency filtered music reduce PTSD symptoms for patients receiving cognitive processing therapy for PTSD?
* Does the addition of frequency filtered music to cognitive processing therapy improve stress physiology (arousal)?
* Does improvement in physiological stress regulation help explain improvements in hyperarousal and PTSD symptoms? Researchers will compare the effects of a frequency filtered classical music playlist to an identical playlist without added filtering. Participants will be randomized to a music playlist.

Participants will:

* Receive 10 daily sessions of cognitive processing therapy
* Listen to 15 minutes of music before their therapy sessions (2.5 hours music listening total).
* Complete clinical interviews and questionnaires before, during, and up to 6 months after therapy.
* Have their physiological arousal monitored during listening and therapy sessions
* Wear a Fitbit device and complete smartphone surveys for 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Meets diagnostic criteria for a) PTSD or b) subthreshold PTSD with hyperarousal (i.e., meets diagnostic threshold for 3 of 4 symptoms, one of which is hyperarousal)
* Ability to move between sitting to standing without assistance
* Ability to attend two weeks of daily in-person therapy sessions at either the Ohio State University or at the Wright-Patterson Air Force Base (WPAFB) Medical Center

Exclusion Criteria:

* Heart condition (such as cardiac arrhythmia) or pacemaker
* An allergy that would prevent wearing adhesive for durations of 2 hours or less
* Insufficient English fluency to fully engage in psychotherapy
* Use of hearing aids
* Current or prior tinnitus (persistent ringing or other noises in ears not caused by an external sound)
* Severe traumatic brain injury
* An ongoing stressor or condition deemed by the investigators to place the participant at risk for injury or a poor outcome (e.g., undergoing disability evaluation, undergoing a medical board evaluation to be medically discharged from the military, pending negative administrative or legal actions).
* Inability to complete the informed consent process due to the acute effects of a medical or psychiatric condition (e.g., intoxication, mania, psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2028-02-14 (Estimated); Study Completion 2028-02-14 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptom Severity (Self Rated) | 1 month after treatment completion
  PTSD symptom severity will be assessed using the PTSD Checklist for DSM 5 (PCL-5). The scale includes 20 items that rate the severity of each symptom using a 5-point scale, with items summed to provide an overall metric of PTSD symptom severity.
PTSD Symptom Severity (Self Rated) | 3 months after treatment completion
  PTSD symptom severity will be assessed using the PTSD Checklist for DSM 5 (PCL-5). The scale includes 20 items that rate the severity of each symptom using a 5-point scale, with items summed to provide an overall metric of PTSD symptom severity.
PTSD Symptom Severity (Self Rated) | 6 months after treatment completion
  PTSD symptom severity will be assessed using the PTSD Checklist for DSM 5 (PCL-5). The scale includes 20 items that rate the severity of each symptom using a 5-point scale, with items summed to provide an overall metric of PTSD symptom severity.

SECONDARY OUTCOMES:
PTSD Symptom Severity (Clinician Rated) | 1 month after treatment completion
  PTSD symptom severity as measured by the Clinician Administered PTSD Scale for DSM-5 Revised (CAPS-5-R)
PTSD Symptom Severity (Clinician Rated) | 3 months after treatment completion
  PTSD symptom severity as measured by the Clinician Administered PTSD Scale for DSM-5 Revised (CAPS-5-R)
PTSD Symptom Severity (Clinician Rated) | 6 months after treatment completion
  PTSD symptom severity as measured by the Clinician Administered PTSD Scale for DSM-5 Revised (CAPS-5-R)
Hyperarousal Symptom Severity (Self Rated) | 1 month after treatment completion
  Hyperarousal symptoms will also be measured using items from the PCL-5. Hyperarousal symptom severity is calculated by summing the 6 Criterion E items of each scale (i.e., items 15-20), such that higher scores indicate more severe hyperarousal.
Hyperarousal Symptom Severity (Self Rated) | 3 months after treatment completion
  Hyperarousal symptoms will also be measured using items from the PCL-5. Hyperarousal symptom severity is calculated by summing the 6 Criterion E items of each scale (i.e., items 15-20), such that higher scores indicate more severe hyperarousal.
Hyperarousal Symptom Severity (Self Rated) | 6 months after treatment completion
  Hyperarousal symptoms will also be measured using items from the PCL-5. Hyperarousal symptom severity is calculated by summing the 6 Criterion E items of each scale (i.e., items 15-20), such that higher scores indicate more severe hyperarousal.
Hyperarousal Symptom Severity (Clinician Rated) | 1 month after treatment completion
  PTSD symptom severity as measured by the Clinician Administered PTSD Scale for DSM-5 Revised (CAPS-5-R) Criterion E
Hyperarousal Symptom Severity (Clinician Rated) | 3 months after treatment completion
  PTSD symptom severity as measured by the Clinician Administered PTSD Scale for DSM-5 Revised (CAPS-5-R) Criterion E
Hyperarousal Symptom Severity (Clinician Rated) | 6 months after treatment completion
  PTSD symptom severity as measured by the Clinician Administered PTSD Scale for DSM-5 Revised (CAPS-5-R) Criterion E
PTSD Diagnosis (Clinician Rated) | 1 month after treatment completion
  PTSD diagnosis as assessed by the Clinician Administered PTSD Scale for DSM-5 Revised (CAPS-5-R)
PTSD Diagnosis (Clinician Rated) | 3 months after treatment completion
  PTSD diagnosis as assessed by the Clinician Administered PTSD Scale for DSM-5 Revised (CAPS-5-R)
PTSD Diagnosis (Clinician Rated) | 6 months after treatment completion
  PTSD diagnosis as assessed by the Clinician Administered PTSD Scale for DSM-5 Revised (CAPS-5-R)
Change in resting parasympathetic activity | Change from 1 week before treatment start to 1 week after treatment completion
  High-frequency heart rate variability during seated rest will be calculated from electrocardigram data using CardioBatch Plus software. Range: 0 - 15 ln(msec). Greater variability indicates greater parasympathetic vagal activity
Change in resting physiological arousal | Change from 1 week before treatment start to 1 week after treatment completion
  Mean heart period during seated rest will be calculated from electrocardigram data. Range: 200-1500 msec. Longer heart period indicates lower physiological arousal.
Change in parasympathetic activity during cognitive stress test | Change from 1 week before treatment start to 1 week after treatment completion
  High-frequency heart rate variability response to a cognitive stress test from resting baseline will be calculated from electrocardigram data using CardioBatch Plus software.
Change in sympathetic activity during cognitive stress test | Change from 1 week before treatment start to 1 week after treatment completion
  Change in rate of skin conductance response firing per minute to a cognitive stress test from resting baseline will be calculated. Faster rate indicates more sympathetic activation.
Change in cardiac physiological arousal during cognitive stress test | Change from 1 week before treatment start to 1 week after treatment completion
  Change in mean heart period to a cognitive stress test from resting baseline will be calculated. Shorter mean heart period indicates greater arousal.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Ohio State University, Columbus, Ohio
  - Wright Patterson Air Force Base Mental Health Center, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Researchers interested in using IPD and/or computer code collected or generated as part of this study may do so by contacting the study PI. Researchers will be asked to complete a Data Use Request Form, which includes contact information, description of the research project for which the data and/or code would be used, specification of which data and/or code would be needed for their proposed project, an approximate time line for their proposed project, and authorship on their proposed project.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication of primary results
Access Criteria: All requests for data and/or code use will be reviewed by the PIs and co-Is and a majority vote will be used to determine whether the request is approved or not. If the request is approved, Dr. Kolacz will inform the requestor, return a signed copy of the completed Data Use Request Form to the requestor, and let the requestor know that written IRB approval of the requestor's proposed study from the requestor's home institution will be required before data and/or code will be shared with the requestor. If a request is approved pending revision to the Data Use Request Form, Dr. Kolacz will work with requestors to revise sections of their Data Use Request Forms in order to obtain approval. If the request is not approved, Dr. Kolacz will inform the requestor and returned a signed copy of the completed Data Use Request Form to the requestor that includes an explanation for the denial.